CLINICAL TRIAL: NCT00390195
Title: Randomized Phase I/II of Rapamycin Analog, RAD001, in Advanced Hepatocellular Carcinoma - With a Pharmacokinetic Study of RAD001
Brief Title: Randomized Phase I/II of RAD001 in Advanced Hepatocellular Carcinoma (HCC)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: Novartis (Industry)
Responsible Party: National Institute of Cancer Research, National Health Research Instiutes, Deputy Director
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001C2453
Record Dates: First submitted 2006-10-17; First posted 2006-10-19 (Estimated); Last update posted 2009-07-02 (Estimated); Status verified 2009-06

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; RAD001; Rapamycin; Randomize; Phase I; Phase II; Pharmacokinetics
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Everolimus

ARMS (2):
- 1. Daily (Experimental): Taking orally the investigational drug daily
  Interventions: Drug: RAD001 (everolimus)
- 2. Weekly (Experimental): Taking orally the investigational drug weekly
  Interventions: Drug: RAD001 (everolimus)

INTERVENTIONS:
Drug: RAD001 (everolimus) — Arm 1: 2.5, 5, 7.5 or 10 mg of RAD001 daily
  Other Names: Certican
  Arms: 1. Daily
Drug: RAD001 (everolimus) — Arm 2: 20, 30, 50 or 70 mg of RAD001 daily
  Other Names: Certican
  Arms: 2. Weekly

SUMMARY:
The mTOR has been examined in hepatocellular carcinomas as well. This pathway is up-regulated in a proportion of hepatocellular carcinoma (HCC) and that rapamycin inhibits cell proliferation and blocks S6K phosphorylation. Inhibition of mTOR had been shown to suppress substantially the liver tumor growth. Nevertheless, inhibition of mTOR was demonstrated to have a clinical response in some cancer types. These reports imply that inhibition of mTOR could be a promising therapeutic strategy in the treatment of HCC. Therefore, we hypothesize that RAD001, a rapamycin analog, can inhibit the mTOR, and subsequently suppress the liver tumor in the treatment of HCC patients.

This study is aimed to investigate the safety, efficacy, pharmacokinetics, pharmacogenetics and feasibility of RAD001 in advanced HCC patients. This study will be a randomized phase I study with dose escalation and subsequently a phase II study of intent to treat, as well as pharmacokinetic, pharmacogenetic and surrogate marker study of RAD001.

DETAILED DESCRIPTION:
Objectives：

1. Primary Objectives

   * Phase I: To assess the maximal tolerated dose (MTD) of once daily and weekly oral RAD001 in patients with advanced HCC of Child-Pugh's class A or B
   * Phase II: To assess the disease control rate of advanced Child-Pugh's class A or B HCC patients receiving the determined MTD of once daily and weekly oral RAD001 in phase I
2. Secondary Objectives

   * Phase I: To investigate the following items in the advanced HCC patients receiving RAD001

     1. Dose-limiting toxicity
     2. Pharmacokinetics study
     3. Pharmacogenetic study
     4. Surrogate marker study on the PTEN, total and Phosphorylated forms of Akt of tumor tissues
     5. Disease control rate
   * Phase II: To investigate the following items in the advanced HCC patients receiving RAD001

     1. Overall survival
     2. Toxicity profile
     3. Pharmacogenetic study
     4. Surrogate marker study on the PTEN, total and Phosphorylated forms of Akt of tumor tissues

Study Design: This study will be a randomized phase I study with dose escalation and subsequently a phase II study of intent to treat, as well as pharmacokinetic, pharmacogenetic and surrogate marker study of RAD001.

Sample Size: Upto 134 patients (Phase I: in cohort of 3-6 to test each dose level and a upto 48 patients to reach the expected MTD, 24 patients in each schedule of treatment arm; Phase II: 18 patients of each schedule at the first stage and 25 patients of each schedule at the second stage).

Study Medication: The RAD001 dose level of daily schedule will be escalated from 2.5, 5.0, 7.5 to 10 mg/day without splitting, with or without food. The RAD001 dose level of weekly schedule will be escalated from 20, 30, 50 to 70 mg/week without splitting. The dose and schedule of RAD001 in the phase II study will be dependent on the result of phase I study. RAD001 will be supplied by Novartis Co.,

Study Conduct: Patients will be enrolled onto a sequence of receiving an oral dose of RAD001. The schedule of RAD001 will be either once daily or once weekly. Throughout the whole phase I and II study, an eligible patient will be randomized into either arm of daily or weekly schedule. In the phase I part, each cohort of dose level will have 3 patients. The dose of oral RAD001 will be initially fixed at 2.5 gm/day in daily schedule arm and at 20 mg/week in weekly schedule arm. One treatment course is defined as 4 weeks of RAD001 therapy. When no patient experiences dose-limiting toxicity (DLT) at certain level, subsequent patients would be randomized to the next dose level. When 1 out of 3 patients developed DLT, 3 additional patients would be treated with the same dose level. Three patients will be further recruited to the next dose level when none of that 3 additional patients experience DLT. No intra-individual dose-escalation will be performed. In the phase II part, Simon's optimal two-stage approach will be used in both daily and weekly schedules. If one responder is observed at the first stage of eighteen patients in either treatment schedule, further twenty-five patients will be accrued.

Therapeutic Assessment：

1. Efficacy assessment:

   * Radiological response: To evaluate the disease control rate (complete response + partial response + stable disease) by computed tomography after every 8 weeks of therapy and according to RECIST guideline.
   * Biological response

     1. To evaluate the change of serum a-fetoprotein level.
     2. To evaluate the change of plasma angiogenic factors levels.
2. Safety Assessment: Toxicity assessment:

   * Evaluation of toxicity will be performed on patient-base.
   * Clinical and laboratory toxicity/symptomatology will be graded according to NCI common toxicity criteria (CTC) version 3.0.
   * Abnormal liver functional tests are common in patients with HCC, only abnormal elevation of ALT will be considered as indicator of hepatotoxicity.
3. Pharmacokinetic, Pharmacogenetic & Surrogate Marker Assessments

   * Pharmacokinetic assessments:

     1. Cmax: peak concentration
     2. tmax: time to achieve peak concentration
     3. Cmin: trough concentration
     4. Cave: average concentration
     5. AUCt: area under curve within a given time
     6. t1/2: elimination half life
   * Pharmacogenetic assessments:

     1. Polymorphic CYP3A4
     2. Polymorphic CYP3A5
     3. Polymorphic P-glycoprotein
   * Surrogate marker assessments:

     1. PTEN
     2. Total and Phosphorylated forms of Akt

Procedures:

1. Screening will be done within 2 weeks before starting treatment, and will include all parameters listed below, (except for pharmacokinetics, AEs/concomitant medications, and toxicity assessments) as well as informed consent, patient eligibility, medical history, a pregnancy test (if indicated), EKG, and urinalysis.
2. During treatment:

   * Physical examination (including vital sign measurements), height, weight, AEs, and toxicity evaluation at the first day of each week during the initial 4 weeks, biweekly at the subsequently 8 weeks and 4-weekly thereafter.
   * Performance status will be assessed on the first day of each treatment course.
   * Investigators/research nurses should monitor patients in each treatment course and should instruct patients regarding the signs and symptoms of RAD001 toxicity as described in the "Information for Patients" section of the RAD001 product labeling.
   * The laboratory tests, hemogram, clinical chemistry will be conducted weekly at the first 4 weeks, biweekly at the subsequent 8 weeks and 4- weekly thereafter.
   * Imaging studies for tumor response will be performed every 2 courses.
   * Patient clinical and biological responses will be noted at the end of the study.

Statistical Analysis: No formal inferential statistical analyses will be performed. Data will be summarized using descriptive statistics (number of patients, mean, median, standard deviation, minimum, and maximum) for continuous variables and using frequency and percentage for discrete variables. For the safety analyses, data will be presented for all patients. An accounting of the study patients by disposition will be tabulated. Demographic data (e.g., age, gender), medical history, cancer history, and other baseline characteristics will be summarized.

1. Safety Evaluation: The general safety and tolerability of RAD001 will be assessed using the following safety endpoints: AEs, routine clinical laboratory evaluations (hemogram, serum chemistry, and urinalysis), physical examination, concomitant medications, and Eastern Cooperative Oncology Group (ECOG) performance status. The grade of AEs at the time of rescue as determined from the NCI-CTC version 3.0.
2. Pharmacokinetic Analysis: Pharmacokinetic parameters will be determined from plasma drug and metabolite concentration curves using non- compartmental approaches. Mean (SD) plasma drug concentration values will be summarized and plotted for each dose group. All parameters described will be summarized with means and standard deviations. The concentration in plasma determined at each sampling time point will be furnished on the original scale for each subject participating in the study. The pharmacokinetic parameters Cmax, Cmin, Cave, and AUC will be analyzed on the logarithmic scale of measurement. The parameters of elimination half- life and tmax will be analyzed on the original scale.
3. Efficacy Analysis: The efficacious parameters will be determined by mean of disease control rate and median of time to tumor progression (TTP) and overall survival (OS) using Kaplan-Meier method. The efficacious parameters will be added with 95% confidence interval. All calculations will be based on the intent-to-treat principle.

ELIGIBILITY:
Inclusion Criteria:

* Patients with measurable, metastatic or locally advanced HCC that are not feasible to have or have failed to prior local therapy (including surgical resection, transarterial chemoembolization and/or alcohol injection) are eligible.
* The diagnosis of HCC should be established either by cyto/histology; or, by characteristic imaging studies (have to including angiography) plus serum level of AFP equal to or more than 400 ng/mL in patients with cirrhosis of the liver and/or chronic viral hepatitis B or C infection.
* Patients must be equal to or more than 20 years of age and equal or less than 75 years of age.
* Patients must have a performance status of ECOG score equal to or less than 2.
* Patients must fulfill all of the following criteria: Child-Pugh's Score equal to or less than 9; serum total bilirubin level is equal to or less than 2.0 mg/dL; serum ALT level (GPT) equal to or less than 3.0 x upper normal limit; platelet are equal to or more than 50,000 / uL; WBC are equal to or more than 3,000 / uL.
* Serum creatinine equal to or less than 2.0 x upper normal limit.
* Life expectancy equal to or more than 12 weeks.
* Signed informed consent.
* Sexually active patients, in conjunction with their partner, must practice birth control during, and for 2 months after therapy.
* Female patients at child-bearing age must have negative pregnancy test.
* No known HIV infection.

Exclusion Criteria:

* Patients with diseases which require concurrent usage of glucocorticosteroid or immunosuppressant agent(s) are not eligible.
* Patients with concomitant active secondary malignancies, except for surgically cured carcinoma in situ of the cervix and basal or adequately treated squamous cell carcinoma of the skin, or disease-free of malignancies < 3 years before the study, are not eligible.
* Patients with active infection are not eligible.
* Patients who received other rapamycin analogs before are not eligible.
* Patients with severe cardiopulmonary diseases (including history of stable, effort-induced or unstable angina pectoris or myocardiac infarction) and other systemic diseases under poor control are not eligible.
* Patients with history of psychiatric disorder are not eligible.
* Patients with brain metastases are not eligible.
* Patients who received surgery, radiotherapy except to bone, chemotherapy, immunotherapy, or other investigational drug within 4 weeks before initiating study are not eligible.
* Patients who are pregnant, breast-feeding or not using appropriate birth control during the course of the study are not eligible.
* Patients with significant concomitant disease that will be aggravated by the investigational drug are not eligible.
* Patients on active treatment with inhibitors or inducers of P-glycoprotein, CYP3A4 and CYP3A5 are not eligible; a minimal of 2 weeks wash-out period will be required after stop such medications.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2006-10; Primary Completion 2010-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose in Phase I | June-2008
Disease control rate in Phase II | Dec-2009

SECONDARY OUTCOMES:
Angiogenic factors | Dec-2009
Pharmacokinetics | Jun-2008
Pharmacogenetics | Dec-2009
Pharmacodynamics | Dec-2009
Overall survival | Jun-2010
Time to tumor progression | Jun-2010
Tumor marker | Dec-2009

CONTACTS AND LOCATIONS:
Overall Officials: Li-Tzong Chen, M.D., Ph.D., Principal Investigator — National Institute of Cancer Research, National Health Research Institutes, Taiwan
Locations (2):
- Taiwan (2):
  - National Cheng Kung University Hospital, Tainan
  - Tri-Service General Hospital, Taipei

REFERENCES:
- [Background] Chan S. Targeting the mammalian target of rapamycin (mTOR): a new approach to treating cancer. Br J Cancer. 2004 Oct 18;91(8):1420-4. doi: 10.1038/sj.bjc.6602162. PMID 15365568
- [Background] Meric-Bernstam F, Mills GB. Mammalian target of rapamycin. Semin Oncol. 2004 Dec;31(6 Suppl 16):10-7; discussion 33. doi: 10.1053/j.seminoncol.2004.10.013. PMID 15799239
- [Background] Bjornsti MA, Houghton PJ. The TOR pathway: a target for cancer therapy. Nat Rev Cancer. 2004 May;4(5):335-48. doi: 10.1038/nrc1362. No abstract available. PMID 15122205
- [Result] Yee KW, Zeng Z, Konopleva M, Verstovsek S, Ravandi F, Ferrajoli A, Thomas D, Wierda W, Apostolidou E, Albitar M, O'Brien S, Andreeff M, Giles FJ. Phase I/II study of the mammalian target of rapamycin inhibitor everolimus (RAD001) in patients with relapsed or refractory hematologic malignancies. Clin Cancer Res. 2006 Sep 1;12(17):5165-73. doi: 10.1158/1078-0432.CCR-06-0764. PMID 16951235
- [Result] Sahin F, Kannangai R, Adegbola O, Wang J, Su G, Torbenson M. mTOR and P70 S6 kinase expression in primary liver neoplasms. Clin Cancer Res. 2004 Dec 15;10(24):8421-5. doi: 10.1158/1078-0432.CCR-04-0941. PMID 15623621
- [Result] Rizell M, Lindner P. Inhibition of mTOR suppresses experimental liver tumours. Anticancer Res. 2005 Mar-Apr;25(2A):789-93. PMID 15868910
- [Derived] Shiah HS, Chen CY, Dai CY, Hsiao CF, Lin YJ, Su WC, Chang JY, Whang-Peng J, Lin PW, Huang JD, Chen LT. Randomised clinical trial: comparison of two everolimus dosing schedules in patients with advanced hepatocellular carcinoma. Aliment Pharmacol Ther. 2013 Jan;37(1):62-73. doi: 10.1111/apt.12132. Epub 2012 Nov 8. PMID 23134470
- [Derived] Treiber G. mTOR inhibitors for hepatocellular cancer: a forward-moving target. Expert Rev Anticancer Ther. 2009 Feb;9(2):247-61. doi: 10.1586/14737140.9.2.247. PMID 19192962